CLINICAL TRIAL: NCT04401631
Title: Analytical Validation of the abioSCOPE Device With an IgE Test Panel: Point-of-Care Precision, Sample Type Comparison and Method Correlation
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor financial has been stopped
Sponsor: Abionic SA (Industry)
Collaborators: NAMSA (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: AB-ALL-3.1
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Allergy; Allergic Asthma; Allergy to Cats; Allergy to House Dust; Allergy to Dog Dander (Finding); Allergy Mold; Allergy Cockroach
Keywords: Allergy; Asthma; Point-of-Care; Immunoassay; In vitro Diagnostic; Total IgE; Specific allergy
MeSH Terms: conditions — Hypersensitivity; Signs and Symptoms; Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interventions: * A minimum of 20 subjects with targeted levels of total IgE are needed to participate in the Operator-to-Operator whole blood study.
  * A minimum of 20 subjects with targeted levels of allergen-specific and total IgE are needed to participate in the capillary whole blood between-run imprecision study in the POL environment.
  * A minimum of 40 subjects with targeted levels of Fel d 1-specific IgE and total IgE are needed to participate in the sample type comparison study. These subjects will be recruited, and their samples analyzed at 1 POL.
  * A minimum of 300 subjects (approximately 100 subjects enrolled and evaluated at each of three sites) and with targeted levels of total IgE are needed to participate in the method comparison study.
  Interventions: Device: Blood Collection

INTERVENTIONS:
Device: Blood Collection — Between-Run Reproducibility K3-EDTA venous whole blood 3 mL 1 venous draw
  Operator-to-operator imprecision (abioSCOPE) K3-EDTA capillary whole blood 0.05 mL/draw; 0.15 mL total 3 finger sticks (3 different fingers)
  Sample type comparison (abioSCOPE) K3-EDTA capillary whole blood, venous serum, venous K3-EDTA plasma 0.35 mL (finger stick), 9 mL of whole blood to get a minimum of 3 mL of serum and 9 mL of whole blood K3-EDTA to get a minimum of 3 mL of plasma 1 finger stick; 1 venous draw into serum tube (9 mL) and 1 venous draw into K3-EDTA plasma tube (9 mL), in total 18 mL
  Method comparison (abioSCOPE and ImmunoCAP/Phadia) K3-EDTA capillary whole blood, venous K3-EDTA plasma 0.05 mL (finger stick), 9 mL of whole blood to get a minimum of 3 ml of plasma 1 finger stick; 1 venous draw into K3-EDTA plasma tube (9 mL tube)

SUMMARY:
This is a multicenter, prospective, observational study to evaluate the analytical performance of the Abionic IgE Multi-Allergen Test Panel on the abioSCOPE® device in a U.S. point-of-care environment within a clinical laboratory operating under a CLIA certificate for tests of moderate complexity. The study will assess point-of-care ('external') precision, sample type comparison and correlation with a reference method (Phadia Laboratory System, ThermoFisher Scientific).

ELIGIBILITY:
Inclusion Criteria:

* Provision and understanding of signed and dated written informed consent by the subject prior to any mandatory study-specific procedures, sample collection, or analysis.
* Male or female, 18 years of age or older.

Exclusion Criteria:

* Subject participating in another study that may influence test results.
* Subject taking any of the following medications: systemic steroids (inhaled or nasal steroids are allowed), anti-cytokines or cytokines, systemic interferon (injection local interferon α for the treatment of HPV is allowed), anti-IgE therapy (approved or investigational) or treated with systemic chemotherapy.
* History of cancer, autoimmune, or immune deficiency disease.
* Suffering from a hematological pathology (coagulation disorder, severe anemia) that could interfere with the blood draw procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * A minimum of 20 subjects with targeted levels of total IgE are needed to participate in the Operator-to-Operator whole blood study.
  * A minimum of 20 subjects with targeted levels of allergen-specific and total IgE are needed to participate in the capillary whole blood between-run imprecision study in the POL environment.
  * A minimum of 40 subjects with targeted levels of Fel d 1-specific IgE and total IgE are needed to participate in the sample type comparison study. These subjects will be recruited, and their samples analyzed at 1 POL.
  * A minimum of 300 subjects (approximately 100 subjects enrolled and evaluated at each of three sites) and with targeted levels of total IgE are needed to participate in the method comparison study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
POC variance components (in a POL environment): | Day 1
  * External Precision Study ('reproducibility study' 'site-to-site precision study'): Demonstrate that the imprecision of K3-EDTA venous plasma using the IVD CAPSULE Allergic Asthma panel on the abioSCOPE device (all 5 allergens/allergen mixes and total IgE) in the hands of trained Healthcare Professionals in a Physician Office Laboratory (POL) is within the expected range of the imprecision established in the clinical laboratory by Laboratory Scientists.
  * Operator-to-Operator imprecision on whole blood: Demonstrate that the between-Operator reproducibility of the total IgE of the IVD CAPSULE Allergic Asthma panel on the abioSCOPE device test results is within the expected range of variability.
  * Between-run reproducibility: Demonstrate that the between-run reproducibility of venous whole blood samples measured with the IVD CAPSULE Allergic Asthma panel on the abioSCOPE device (all 5 allergens/allergen mixes and total IgE) is within the expected range of variability.
Sample type comparison: | Day 1
  Demonstrate that the IVD CAPSULE Allergic Asthma panel on the abioSCOPE device test results obtained from capillary whole blood correlates well with values obtained from K3-EDTA anticoagulated venous plasma and serum samples.
Method comparison | Day 1
  Demonstrate that test results obtained with the total IgE test of the IVD CAPSULE Allergic Asthma panel on the abioSCOPE device correlates with total IgE test results from the reference method (Phadia Laboratory System, ThermoFisher Scientific).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - George Washington University, Washington DC, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Baltimore, Maryland
  - The Bernstein Clinical Research Center Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided